CLINICAL TRIAL: NCT06336889
Title: Pelvic Angioembolization: A Prospective Multi-Institutional Study (Data From All Campuses Will be Used)
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 092.TRA.2018.D
Record Dates: First submitted 2022-04-27; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pelvic Angioembolization — Embolization is performed by placing a small catheter inside the blood vessels that supply the area that is bleeding. Carefully navigating the catheter, under image guidance, to the safest and farthest point, a variety of different materials can then be used to block the bleeding vessels.

SUMMARY:
The investigator's propose a multicenter prospective observational study to investigate the use of embolization in patients with negative angiogram and to ascertain the optimal level of treatment when the angiogram is positive; non-selective vs. selective embolization.

DETAILED DESCRIPTION:
The investigator's propose a multicenter prospective observational study to investigate the use of embolization in patients with negative angiogram and to ascertain the optimal level of treatment when the angiogram is positive; non-selective vs. selective embolization. The investigator's will divide patients into groups based on positive or negative angiogram. Within each group the investigator's will compare those embolized and level of embolization. All blunt trauma patients undergoing angiography for pelvic fracture associated hemorrhage will be eligible for the study. Demographic, physiologic, operative, and post-operative data will be collected including blood product resuscitation, classification and management of pelvic fracture, associated injuries, angiographic details, complications, outcomes and overall injury burden. The study population will be stratified based on presence of arterial hemorrhage on initial angiogram (positive or negative angiogram) and then further stratified based on performance of embolization. NSE will be defined as embolization of the main internal iliac artery, either unilaterally or bilaterally and SE as any embolization distal to the main internal iliac artery. Bivariable and multivariable analyses will be performed to determine differences in pelvic hemorrhage as measured by transfusion necessity and quantity of products required, complications and to identify independent risk factors for outcome variables. A power analysis was performed based off of thromboembolic complication difference in selective vs. non selective embolization and then again with blood transfusion requirement difference in embolized vs. not embolized for those who have no evidence of arterial bleeding on angiogram (IE the two questions the investigator's are trying to answer).The investigator's plan to complete the data collection and analysis by 1/1/2019.

ELIGIBILITY:
Inclusion Criteria:

* • All blunt trauma patients undergoing angiography for pelvic fracture associated hemorrhage

Exclusion Criteria:

* • Pregnant patients

  * Patients < 18 years old
  * Patients undergoing angiography greater than 24 hours from arrival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator will ensure that this study is conducted in full conformity with the principles set forth in The Belmont Report: Ethical Principles and Guidelines for the Protection of Human Subjects of Research, as drafted by the US National Commission for the Protection of Human Subjects of Biomedical and Behavioral Research (April 18, 1979) and codified in 45 CFR Part 46 and/or the ICH E6. If the study is conducted at international sites, the statement could be as above and/or could reference compliance with the Declaration of Helsinki, CIOMS, International Ethical Guidelines for Biomedical Research Involving Human Subjects (2002), or another country's ethical policy statement, whichever provides the most protection to human subjects.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Mortality outcome | 2018-2019
  Dead or Alive
transfusion requirements | 2018-2019
  transfusion requirements
thromboembolic events | 2018-2019
  thromboembolic events

SECONDARY OUTCOMES:
Patient demographics(age, sex) | 2018-2019
  Patient demographics

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Burris, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided